CLINICAL TRIAL: NCT03374501
Title: Determination of the Glycemic and Insulinemic Index Values of Soft Drink and Two Test Meals Containing Soft Drink Consumed With Sugardown™
Brief Title: Determination of the GI and II Values of Soft Drink and Soft Drink With Sugardown™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: PAZ320-004
Record Dates: First submitted 2017-12-12; First posted 2017-12-15 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Postprandial Hyperglycemia
Keywords: Sugardown™; Galactomannan; Postprandial blood glucose; Insulin
MeSH Terms: conditions — Hyperglycemia; Insulin Resistance | interventions — PAZ320; Carbonated Beverages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2 tablets Sugardown™ (Experimental): Repeated-measures, open cross-over design: 10 subjects consumed three different test meals comprising of soft drink consumed with 2 tablets of Sugardown™
  Interventions: Dietary Supplement: Sugardown™
- 4 tablets Sugardown™ (Experimental): Repeated-measures, open cross-over design: 10 subjects consumed three different test meals comprising of soft drink consumed with 4 tablets of Sugardown™
  Interventions: Dietary Supplement: Sugardown™
- Soft drink (Placebo Comparator): Repeated-measures, open cross-over design: 10 subjects consumed three different test meals comprising of soft drink
  Interventions: Dietary Supplement: Soft drink

INTERVENTIONS:
Dietary Supplement: Sugardown™ — Test food #2: 495.0 g Sprite™ soft drink plus 2 Sugardown™ tablet consumed with 250 mL water (repeated twice) Test food #3: 495.0 g Sprite™ soft drink plus 4 Sugardown™ tablet consumed with 250 mL water (repeated twice)
  Other Names: BTI320; PAZ320
  Arms: 2 tablets Sugardown™; 4 tablets Sugardown™
Dietary Supplement: Soft drink — Test food #1: 495.0 g Sprite™ soft drink consumed with 250 mL water (repeated twice)
  Other Names: Sprite™
  Arms: Soft drink

SUMMARY:
This study was a partly controlled laboratory-based study comparing the glycemic and insulinemic indices of 3 test meals containing soft drink alone or with SUGARDOWN™ (Galactomannan) in overweight adults.

DETAILED DESCRIPTION:
STUDY SUMMARY This study was a partly controlled, laboratory-based study comparing the short-term postprandial glucose and insulin responses produced by three test meals containing soft drink consumed alone or with SUGARDOWN™, relative to the responses produced by an equal-carbohydrate portion of glucose solution (the reference food). The study used a repeated measures design, such that every subject consumed the reference food and each test food on two separate occasions, completing a total of eight separate test sessions. Each subject completed their test sessions on separate weekday mornings at a similar time each day, as close as possible to the time they would normally eat breakfast.

SUBJECTS Ten healthy, non-smoking, overweight or obese subjects (6 females and 4 males) voluntarily participated in this study. The mean ± SD age of the subjects was 32.4 ± 10.9 yr (range: 18.7 - 55.6 yr), and their mean ± body mass index value was 27.4 ± 2.6 kg/m2 (range: 25.3 - 32.3 kg/m2).

Volunteers were given detailed written and verbal information about all of the study's inclusion criteria and experimental procedures. If the volunteers decided that they would like to participate in the study, they were asked to come to the research centre on another morning, where they completed a detailed screening questionnaire that assessed their current health status and medical history. In order to participate in the study, the volunteers had to meet the inclusion criteria. All suitable volunteers that were invited to participate in the study were required to sign a detailed subject information sheet and a consent form before commencing any experimental procedures.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-65 years.
* Non-smoker.
* Stable body weight within the overweight weight range for their height (BMI values 25 kg/m2 for Causcasian individuals and >23 kg/m2 for Asian individuals).
* Normal dietary habits; not dieting or eating in an overly restrictive fashion in the past 3 months.
* A regular pattern of low to moderate physical activity.
* Able to fast for ≥ 10 hours the night before each test session.
* Able to refrain from eating a legume-based evening meal or drinking alcohol the day before each test session.
* Finds the test foods suitable for consumption within 12 minutes.
* Not taking any treatment for anorexia, weight loss, or any form of treatment or medication likely to interfere with metabolism or dietary habits.
* Signed the informed consent form for the study.

Exclusion Criteria:

* Currently following a restrictive diet (low-calorie, low-carbohydrate, vegan).
* Any clinically significant physical or mental illness.
* Suffering from a food allergy or serious food intolerance.
* Regularly taking prescription medication other than standard contraceptive medication.
* Females who are currently pregnant, breast-feeding, trying to become pregnant or not using an acceptable contraceptive.
* Participating in another clinical trial or participated in another clinical trial within the two weeks.
* Undergoing general anaesthesia in the month prior to inclusion.
* Subject in a situation, which in the investigator's opinion could interfere with optimal participation in the present study or could constitute a special risk for the subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Glycemic index of the three test meals. | 2 days
  Blood samples were collected into a micro-centrifuge tube containing the anticoagulant, heparin sodium salt. Plasma glucose concentrations were measured in duplicate using a spectrophotometric centrifugal analyser employing the glucose hexokinase/glucose-6-phosphate dehydrogenase enzymatic assay.

SECONDARY OUTCOMES:
Insulinemic index of the three test meals. | 2 days
  Each blood sample was collected into a micro-centrifuge tube containing the anticoagulant. Plasma insulin concentrations were measured using a solid phase antibody-coated tube radioimmunoassay kit.

CONTACTS AND LOCATIONS:
Overall Officials: Jennie Brand-Miller, Principal Investigator — School of Molecular Bioscience, University of Syndey, Australia